CLINICAL TRIAL: NCT04875364
Title: Do Endotypes Predict Response and Sequelae in OSA Patients
Acronym: ExPRESSION
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Atul Malhotra, Professor, Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201432
Record Dates: First submitted 2021-04-27; First posted 2021-05-06 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Obstructive Sleep Apnea; Sleep Apnea; Sleep Apnea, Obstructive; Sleep; Sleep Disorder
Keywords: sleep; sleep apnea; OSA; obstructive sleep apnea; lunesta; cpap; endotype; Eszopiclone
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Sleep Wake Disorders; Microcephaly, Primary Autosomal Recessive, 6 | interventions — Eszopiclone; Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Early PAP Start (Experimental): After two initial baseline overnight studies, and two experimental overnight studies during which subjects will receive Eszopiclone (2mg before bedtime) or oxygen (4L/min via nasal cannula for the duration of the time in bed) in random order, subjects will be set up with a loaner CPAP for 8 weeks to initiate therapy right away.
  Interventions: Drug: Eszopiclone; Other: Supplemental Oxygen; Device: Continuous Positive Airway Pressure (CPAP)
- Usual PAP Start (Experimental): After two initial baseline overnight studies, and two experimental overnight studies during which subjects will receive Eszopiclone (2mg before bedtime) or oxygen (4L/min via nasal cannula for the duration of the time in bed) in random order, subjects will remain untreated until they are set up with their clinically prescribed CPAP (typically takes about 8 weeks).
  Interventions: Drug: Eszopiclone; Other: Supplemental Oxygen

INTERVENTIONS:
Drug: Eszopiclone — 2mg of Eszopiclone just before going to sleep.
  Other Names: Lunesta
Other: Supplemental Oxygen — Constant oxygen flow at 4 Liters per minutes for the duration of time in bed via nasal cannula.
Device: Continuous Positive Airway Pressure (CPAP) — A standard CPAP device will be provided using the settings as prescribed by the treating physician.
  Arms: Early PAP Start

SUMMARY:
This study will investigate why some people have Obstructive Sleep Apnea (OSA) and how the underlying cause may relate to OSA manifestations (including sleepiness and high blood pressure) and response to different therapeutic approaches (ie CPAP, eszopiclone, and supplemental oxygen). Understanding why someone has OSA could affect how best to treat that individual, but may also have an impact on what problems the disease might cause.

ELIGIBILITY:
Inclusion Criteria:

* Ages 21-65 years old
* Men and women with a physician diagnosis of OSA (or strongly suspected to have sleep apnea - * see below)
* BMI 20 - 35 kg/m2

Exclusion Criteria:

* Pregnancy (current or planned)
* Nursing
* Inability to provide self-consent or complete study procedures, such as questionnaires that are only available/validated in English.
* Already on effective therapy and adherent to treatment for OSA
* Other known untreated sleep fragmenting disorder, such as periodic limb movement disorder, or narcolepsy
* Circadian rhythm disorder
* Unrevascularized coronary artery disease, angina, prior heart attack or stroke, congestive heart failure
* Uncontrolled hypertension (systolic blood pressure >160, diastolic blood pressure >95)
* Chronic lung disease requiring the use of supplemental oxygen, or with evidence of hypercapnia due to obstructive lung disease.
* Presence of tracheostomy
* Hospitalization within the past 90 days
* Prior peptic ulcer disease, esophageal varices, or gastrointestinal bleeding (< 5 years)
* Prior gastric bypass surgery
* Chronic liver disease or end-stage kidney disease
* Active cancer
* Allergy to any of the study drug
* Regular use of medications known to affect control of breathing (opioids, sedatives/hypnotics including benzodiazepines, theophylline)
* Chronically using study drug (Eszopiclone)
* Active illicit substance use
* Alcohol use of >1 standard drink/night for women or >2 standard drinks/night for men nightly alcohol use
* Active smoking or vaping within the past 6 months
* Psychiatric disease, other than controlled depression/anxiety
* Prisoners

  * Subjects who are strongly suspected to have sleep apnea will be offered an overnight home sleep apnea test (HSAT) to verify OSA diagnosis.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Psychomotor Vigilance Test | 8 weeks
  A 10-minutes, computerized reaction test asking subject to press a button every time a prompt appears. Faster times indicate better reactions and higher alertness.
Endothelial Dysfunction | 8 weeks
  Using a device called EndoPAT for a non-invasive bloodflow measure before, during, and after 5-minutes of occlusion to one arm. Differences in EndoPAT results will be compared between treatments.

SECONDARY OUTCOMES:
Neurocognitive Assessment: NIH Toolbox | 8 weeks
  This battery yields three composite scores: overall cognitive function, crystallized cognition and fluid cognition. The two tests of "crystallized cognition" are less sensitive to acquired brain dysfunction and reflect past learning experiences (Oral Reading Recognition and Picture Vocabulary). The five tests of "fluid cognition" assess multiple cognitive domains that are vulnerable to acquired brain dysfunction (i.e., Picture Sequence Memory Task = episodic memory, Dimensional Change Card Sort Task = executive function/flexibility, Pattern Comparison Task = processing speed, Flanker Inhibitory Control and Attention Task = executive function/inhibitory control, and List Sorting Task = working memory).
Epworth Sleepiness Scale (ESS) | 8 weeks
  A self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP), or their 'daytime sleepiness'.
Pittsburgh Sleep Quality Index (PSQI) | 8 weeks
  A 19-item, self-rated questionnaire designed to measure sleep quality and disturbance over the past month. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.
Insomnia Severity Index (ISI) | 8 weeks
  A 7-item self-report form to assess insomnia severity. Total score categories: 0-7 = No clinically significant insomnia, 8-14 = Subthreshold insomnia, 15-21 = Clinical insomnia (moderate severity), 22-28 = Clinical insomnia (severe).
Richard's Campbell Sleep Questionnaire (RCSQ) | 8 weeks
  A five-item self-report questionnaire that is used in order to assess perceived sleep depth, sleep latency (time to fall asleep), and number of awakenings, as well as sleep efficiency and quality. Each item is scored on a visual analog scale ranging from 0 mm to 100 mm, with higher scores representing better sleep. The mean score of the five items is known as the total score and represents the overall perception of sleep.
Functional Assessment of Chronic Illness Therapy Fatigue Scale (FACIT-F) | 8 weeks
  A 40-item questionnaire to assesses self-reported fatigue and its impact upon daily activities and function. The score ranges from 0 to 160 with greater values indicating better quality of life.
Beck Depression Index-II | 8 weeks
  The questionnaire assesses mental health (i.e. depression). Each of the 21 items are given weighted values corresponding to a symptom of depression and summed to give a single score. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
SF-36 Item Health Survey (SF-36) | 8 weeks
  A set of 36 generic, coherent, and easily administered quality-of-life measures. Scoring consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Brief Pain Inventory (Short Form) | 8 weeks
  A 9 item self-administered questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning. The patient is asked to rate their worst, least, average, and current pain intensity, list current treatments and their perceived effectiveness, and rate the degree that pain interferes with general activity, mood, walking ability, normal work, relations with other persons, sleep, and enjoyment of life on a 10 point scale with 10 being the most pain.
PROMIS (Patient-Reported Outcomes Measurement Information System) pain intensity | 8 weeks
  A self-reported form to assess how much pain a person is feeling.
Systolic Blood Pressure | 8 weeks
  Measured at rest following standard guidelines.
Diastolic Blood Pressure | 8 weeks
  Measured at rest following standard guidelines.
Patient's Assessment of Own Function Inventory (PAOF) questionnaire | 8 weeks
  A subjective measure of cognitive function that asks participants to rate how often they experience difficulty in four areas: memory, language/communication, sensory-motor ability, and executive function with response options from 0 ("almost never") to 5 ("almost always").
PROMIS (Patient-Reported Outcomes Measurement Information System) pain interference | 8 weeks
  A self-reported measure the self-reported consequences of pain on relevant aspects of a person's life and may include the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities.

CONTACTS AND LOCATIONS:
Overall Officials: Atul Malhotra, MD, Principal Investigator — Professor, Medicine; Christopher Schmickl, Principal Investigator — Postdoc Fellow, Medicine
Locations (1):
- Altman Clinical and Translational Research Institute Building, La Jolla, California, United States